CLINICAL TRIAL: NCT04771728
Title: Department of Obstetrics and Gynecology, Peking University Shenzhen Hospital
Brief Title: A Prospective, Randomized Controlled Study of the Probiotics as Adjuvant Treatment for Bacterial Vaginosis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University Shenzhen Hospital (Other)
Collaborators: BGI, China (Other)
Responsible Party: Principal Investigator, Shangrong Fan, Professor of Dept of Obstetrics and Gynecology, Peking University Shenzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUshenzhenH2020-0310
Record Dates: First submitted 2020-09-28; First posted 2021-02-25 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metronidazole vaginal (Active Comparator): Metronidazole vaginal suppositories (200 mg,2 capsules per day,7 days )
  Interventions: Drug: Metronidazole vaginal suppositories
- Metronidazole vagianl and Probiotics(Umeta-mimi) (Experimental): Metronidazole:Metronidazole vaginal suppositories (200 mg,2 capsules per day,7 days ) Probiotics:Oral Umeta-mimi( 5×109cfu per day,30 days）
  Interventions: Drug: Metronidazole vaginal suppositories and Probiotics(Umeta-mimi)

INTERVENTIONS:
Drug: Metronidazole vaginal suppositories — Metronidazole vaginal suppositories (200 mg,2 capsules per day,7 days )
  Arms: Metronidazole vaginal
Drug: Metronidazole vaginal suppositories and Probiotics(Umeta-mimi) — Metronidazole vaginal suppositories (200 mg,2 capsules per day,7 days ) and Oral pobiotics(Umeta-mimi,5×109cfu per day,30 days）
  Other Names: Metronidazole vaginal suppositories adn Probiotics(Umeta-mimi）
  Arms: Metronidazole vagianl and Probiotics(Umeta-mimi)

SUMMARY:
The investigators are trying to determine if oral Probiotics(Umeta-mimi,30 days) with Metronidazole vaginal suppositories (7 days) is better than using Metronidazole vaginal suppositories(7 days) only in preventing the recurrence of bacterial vaginosis

DETAILED DESCRIPTION:
Studies have shown that oral Probiotics(Umeta-mimi) can significantly promote the recovery of vaginal flora mainly because intestinal microbiota can migrate and affect vaginal microecology. This project aims to evaluate the efficacy of oral Probiotics(Umeta-mimi,30 days) with Metronidazole vaginal suppositories(7 days) in the treatment of bacterial vaginosis (BV) and to explore the correlation between vaginal flora and fecal flora by detecting the metagenomics of vaginal secretions and intestinal feces at the time of baseline phase,14 days after treatment， the first month after treatment, 5-7 days after third menstruation after treatment and 5-7 days after sixth menstruation after treatment

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 55 years old, with history of sexual activity,
2. Amsel criterion for diagnosing BV
3. Sign informed consent

Exclusion Criteria:

1. History of systemic organic diseases or psychiatric diseases
2. Planning for or during pregnancy, lactation, menstruation
3. within 5 days of onset of the disease, any antibiotics has been used
4. Long-term use of contraceptives or immunosuppressant
5. Anaphylactic constitution or allergic to known ingredients of research drugs
6. No same fixed partner (RSP) before and after treatment

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Cure rate of BV | 14 days after treatment
  Assessments with different Units of Measure:clinical symptoms such as itching or burning; "fishy" smell; homogeneous thin vaginal discharge;Nugent score; pH>4.5; clue cell.

SECONDARY OUTCOMES:
Recurrence of BV | The first month after treatment
  Nugent score
Recurrence of BV | 5-7 days after third menstruation after treatment
  Nugent score
Recurrence of BV | 5-7 days after sixth menstruation after treatment
  Nugent score

CONTACTS AND LOCATIONS:
Overall Officials: Ruifang Wu, M.D., Study Director — Dept of Obstetrics and Gynecology,Peking University Shenzhen Hospital
Locations (1):
- Peking University Shenzhen Hosptal, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qi F, Fan S, Fang C, Ge L, Lyu J, Huang Z, Zhao S, Zou Y, Huang L, Liu X, Liang Y, Zhang Y, Zhong Y, Zhang H, Xiao L, Zhang X. Orally administrated Lactobacillus gasseri TM13 and Lactobacillus crispatus LG55 can restore the vaginal health of patients recovering from bacterial vaginosis. Front Immunol. 2023 Jul 27;14:1125239. doi: 10.3389/fimmu.2023.1125239. eCollection 2023. PMID 37575226